CLINICAL TRIAL: NCT01894841
Title: Veterans Coping Long-Term With Suicide
Brief Title: Veterans Coping Long-term With Active Suicide
Acronym: CLASP-VA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Butler Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IIR 13-026
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-01

CONDITIONS: Suicide
Keywords: depression; prevention; Veterans health
MeSH Terms: conditions — Suicide; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CLASP Intervention (Experimental): A 6 month adjunctive intervention consisting of 3 individual meetings, one family session, and 11 brief phone contacts with patient and identified significant other.
  Interventions: Behavioral: Coping Long Term with Active Suicide (CLASP); Other: Safety Assessment and Follow Up Evaluation
- Safety Assessment and follow up Evaluation (Other): Treatment as usual plus enhanced monitoring.
  Interventions: Other: Safety Assessment and Follow Up Evaluation

INTERVENTIONS:
Behavioral: Coping Long Term with Active Suicide (CLASP) — 6 month behavioral telephone-based intervention. Calls assess risk, problem solve any immediate issues, and case management
  Arms: CLASP Intervention
Other: Safety Assessment and Follow Up Evaluation — enhanced risk monitoring with full assessment protocol at 3, 6, 9, and 12 month follow up. Results sent as a note to the patient's VA mental health provider

SUMMARY:
The proposed study seeks to test the efficacy of an intervention to reduce suicide behaviors in Veterans. The Veterans Coping Long Term with Active Suicide Program (CLASP-VA) is an innovative, telephone-based intervention that combines elements of individual therapy, case management, and significant other/family therapy and is designed to be integrated into a VA system.

DETAILED DESCRIPTION:
Suicide is a leading cause of death for military personnel, and for the first time in recorded history, rates of military suicides are exceeding civilian rates. Despite public and patient health costs associated with suicidal ideation and behavior, existing efforts haven't appreciably reduced rates of suicidal behavior in the military. Consequently, finding novel, efficacious, and acceptable methods to reduce suicide behaviors is imperative. The Veteran's Coping Long Term with Active Suicide Program (CLASP-VA) is a unique suicide reduction intervention that directly targets high-risk patients at the time of hospital discharge. It is one of the few empirically-developed and promising interventions (e.g., strong pilot data) for individuals hospitalized for suicide behavior.

The primary objective of this study is to test the efficacy of the CLASP intervention compared to a treatment as usual plus Safety Assessment and Follow-up Evaluation (SAFE) control condition. Efficacy will be determined by primary outcomes including: number of attempts, number of re-hospitalizations, severity, and chronicity of suicidal ideation. A secondary objective is identifying the types of patients who receive the most benefit from the CLASP-VA intervention.

ELIGIBILITY:
Inclusion Criteria:

* suicide attempt or suicidal ideation with any methods, plan, and/or intent to make a suicide attempt within 1 week of hospitalization
* age greater than 18
* have a telephone
* ability to speak, read, and understand spoken English sufficiently well to complete the procedures of the study

Exclusion Criteria:

* long-term psychiatric disorder
* diagnosis of borderline personality disorder
* cognitive impairment which would interfere with adequate participation in the project (MMSE <20)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2014-02-24 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Marie Primack, PhD MA, Principal Investigator — Providence VA Medical Center, Providence, RI
Locations (1):
- Providence VA Medical Center, Providence, RI, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Primack JM, Thompson MF, Peters A, Quinn M, Kelsey M, Miller IW, Bozzay M. Suicide Characteristics of Veterans Hospitalized for Suicide Ideation or Attempt. Mil Med. 2023 Nov 3;188(11-12):e3371-e3376. doi: 10.1093/milmed/usad196. PMID 37294816

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Providence VA Medical center psychiatric inpatient unit
Pre-assignment Details: One hundred and seven participants completed baseline assessments and were found to be eligible for the study. Two participants were lost prior to randomization since they could not be contacted by research staff.
Groups:
- CLASP Intervention: The Coping Long Term with Active Suicide is a 6 month adjunctive intervention consisting of 3 individual meetings, one family session, and 11 brief phone contacts with patient and identified significant other.
- Safety Assessment and Follow up Evaluation: Treatment as usual plus enhanced monitoring condition consisting of assessment and medical record notes sent to mental health providers.
  Coping Long Term with Active Suicide: an intervention to reduce suicide behavior in Veterans recently hospitalized for suicide attempt or ideation with intent.
Period: Overall Study
Arm/Group | CLASP Intervention | Safety Assessment and Follow up Evaluation
Started | 52 | 53
Completed | 34 | 44
Not Completed | 18 | 9
Not completed — Withdrawal by Subject | 9 | 4
Not completed — Withdrawn by investigator | 2 | 2
Not completed — Lost to Follow-up | 7 | 3

BASELINE CHARACTERISTICS:
Population: 2 participants completed screening and were enrolled but then were lost to contact prior to completing baseline measures.
Groups:
- CLASP Intervention + Enhanced Monitoring: A 6 month adjunctive intervention consisting of 3 individual meetings, one family session, and 11 brief phone contacts with patient and identified significant other.
  Plus
  Enhanced monitoring consisting of assessment and medical record notes sent to mental health providers.
- Safety Assessment and Follow up Evaluation + TAU: Treatment as usual plus enhanced monitoring condition consisting of assessment and medical record notes sent to mental health providers.
- Total: Total of all reporting groups
Arm/Group | CLASP Intervention + Enhanced Monitoring | Safety Assessment and Follow up Evaluation + TAU | Total
Number analyzed (Participants) | 52 | 53 | 105
Age, Categorical [Count of Participants; unit: Participants] — Demographics survey. Item asked for age of participant at the start of the study. Population: 2 participants were withdrawn from the study after enrollment and randomization prior to completing the baseline assessment.
  Participants
    number analyzed (Participants) | 50 | 53 | 103
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 48 | 47 | 95
    >=65 years | 2 | 6 | 8
Age, Continuous [Mean (Full Range); unit: years] — Population: 2 participants were withdrawn from the study after enrollment and randomization prior to completing the baseline assessment.
  years
    number analyzed (Participants) | 50 | 53 | 103
    (all) | 46.56 [21 to 73] | 48.85 [24 to 83] | 47.705 [21 to 83]
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 2 participants were withdrawn from the study after enrollment and randomization prior to completing the baseline assessment.
  years
    number analyzed (Participants) | 50 | 53 | 103
    (all) | 46.56 (14.07) | 48.85 (14.76) | 47.74 (14.40)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 participants were withdrawn from the study after enrollment and randomization prior to completing the baseline assessment.
  Participants
    number analyzed (Participants) | 50 | 53 | 103
    Female | 4 | 4 | 8
    Male | 46 | 49 | 95
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 2 participants in the CLASP condition failed to complete baseline measures.
  Participants
    number analyzed (Participants) | 50 | 53 | 103
    American Indian or Alaska Native | 0 | 2 | 2
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 4 | 5
    White | 46 | 42 | 88
    More than one race | 1 | 3 | 4
    Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52 | 53 | 105
Beck Hopelessness Scale [Mean (Standard Deviation); unit: units on a scale] — The Beck Hopelessness Scale was used to measure changes in hopelessness from baseline to 12-month followup. Items are dichotomous (0: False and 1: True), with a total score ranging from 0-20. Higher scores indicate greater hopelessness. Population: In the CLASP condition, 2 participants completed screening and were enrolled but then were lost to contact prior to completing baseline measures. An additional 2 failed to complete the full BHI
  2 participants in the SAFE condition did not complete the BHI
  units on a scale
    number analyzed (Participants) | 48 | 51 | 99
    (all) | 12.98 (5.69) | 12.96 (5.53) | 12.97 (5.58)
Columbia Suicide Severity Rating Scale -Ideation [Mean (Standard Deviation); unit: units on a scale] — Intensity of ideation was measured using the Columbia Scale for Suicide Ideation intensity of ideation item. Item responses range from 1 (wish to be dead) to 5 (active suicidal ideation with specific plan and intent), with higher scores indicating more severe ideation. Population: 2 participants completed screening and were enrolled but then were lost to contact prior to completing baseline measures.
  units on a scale
    number analyzed (Participants) | 50 | 53 | 103
    (all) | 4.28 (.730) | 4.26 (.836) | 4.27 (.782)
Columbia Suicide Severity Rating Scale - Attempt Behavior [Mean (Standard Deviation); unit: Suicide attempts] — Items measuring attempt behavior (number of Actual Attempts, number of Aborted Attempts, number of Interrupted Attempts) From the Columbia Suicide Severity Rating Scale were summed to create a composite variable indexing attempt behavior. Higher scores indicate more attempt behavior. Population: 2 participants completed screening and were enrolled but then were lost to contact prior to completing baseline measures.
  Suicide attempts
    number analyzed (Participants) | 50 | 53 | 103
    (all) | 1.40 (1.76) | 1.55 (2.06) | 1.48 (1.92)
WHODAS [Mean (Standard Deviation); unit: units on a scale] — The World Health Organization Disability Assessment Schedule (WHODAS II) is a validated, self-reported instrument assessing current impairment in functioning. Possible scores for each item range from 1 (None) to 5 (Extreme or cannot do). We calculated an Average Global Score for inclusion in analyses by dividing the total score by the number of items included in the measure (possible range of 1-5). Higher scores indicate greater impairment in functioning. Population: 2 participants in CLASP condition were lost prior to baseline completion and 2 additional participants failed to complete the WHODAS
  3 participants in the control condition failed to complete the full WHODAS
  units on a scale
    number analyzed (Participants) | 48 | 50 | 98
    (all) | 93.02 (21.84) | 92.78 (23.67) | 92.90 (22.69)
Brief Symptom Inventory [Mean (Standard Deviation); unit: units on a scale] — The Brief Symptom Inventory is a validated, self-reported instrument assessing current psychiatric symptomatology. Possible scores for each item range from 0 (not at all) to 4 (extremely), and total scores are represented by a Global Severity Index (range 0 to 212). Higher scores indicate greater psychological distress. Population: 2 participants in the CLASp condition were lost prior to completing baseline measures.
  In the SAFE condition, 1 participant had missing data on the BSI
  units on a scale
    number analyzed (Participants) | 50 | 52 | 102
    (all) | 2.02 (.67) | 1.99 (.68) | 2.00 (.68)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Columbia Suicide Severity Rating Scale (C-SSRS) - Behavior
Description: Items measuring attempt behavior (number of Actual Attempts, number of Aborted Attempts, number of Interrupted Attempts) From the Columbia Suicide Severity Rating Scale were summed to create a composite variable indexing attempt behavior. Higher scores indicate more attempt behavior. We log transformed this variable at all time points to meet assumptions of normality.
Time Frame: baseline, 3, 6, 9, & 12 month post-hospitalization
Population: The sample sizes used in this analysis are smaller than the full samples recruited per group because of dropout from baseline to 1 year followup.
Measure: Mean (Standard Deviation); unit: log(attempts)
Arm/Group | CLASP Intervention | Safety Assessment and Follow up Evaluation
Number analyzed (Participants) | 25 | 34
log(attempts)
  Baseline | 0.13 (0.16) | 0.18 (0.21)
  3 Month Followup | 0.14 (0.30) | 0.05 (0.16)
  6 Month Followup | 0.06 (0.15) | 0.01 (0.08)
  9 Month Followup | 0.09 (0.22) | 0.03 (0.11)
  12 Month Followup | 0.06 (0.17) | 0.03 (0.11)
Statistical Analysis 1: Comparison: CLASP Intervention vs Safety Assessment and Follow up Evaluation; Test type: Superiority; p = .13, RMANOVA — Adjusted for change in depression from baseline to 1yr (measured via QIDS); Partial eta squared = .03

2. Secondary Outcome: Changes in Beck Hopelessness Scale
Description: The Beck Hopelessness Scale was used to measure changes in hopelessness from baseline to 12-month followup. Items are dichotomous (0: False and 1: True), with a total score ranging from 0-20. Higher scores indicate greater hopelessness.
Time Frame: Baseline, 3, 6, 9, & 12 month follow up
Population: 2 participants from the CLASP condition were withdrawn from the study after enrollment and randomization prior to completing the baseline assessment. Number of participants analyzed is smaller per group due to dropout from baseline to 12 month follow-up and missing data for some time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CLASP Intervention | Safety Assessment and Follow up Evaluation
Number analyzed (Participants) | 17 | 29
score on a scale
  Baseline | 13.65 (5.62) | 13.21 (5.16)
  3 Month Followup | 9.12 (6.59) | 9.28 (7.32)
  6 Month Followup | 10.06 (7.50) | 9.28 (6.41)
  9 Month Followup | 8.65 (7.13) | 7.31 (6.50)
  12 Month Followup | 9.00 (6.78) | 7.58 (6.72)
Statistical Analysis 1: Comparison: CLASP Intervention vs Safety Assessment and Follow up Evaluation; Test type: Superiority; p = .79, RMANOVA; Adjusted for change in depression from baseline to 1yr (measured via QIDS); Partial eta squared = .01

3. Secondary Outcome: Brief Symptom Inventory
Description: The Brief Symptom Inventory is a validated, self-reported instrument assessing current psychiatric symptomatology. Possible scores for each item range from 0 (not at all) to 4 (extremely), and total scores are represented by a Global Severity Index (range 0 to 212).Higher scores indicate greater psychological distress.
Time Frame: Baseline, 3, 6, 9, & 12 month follow up
Population: There are fewer subjects in this analysis than were recruited for both groups at baseline due to dropout across timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Safety Assessment and Follow up Evaluation: Treatment as usual plus enhanced monitoring condition consisting of assessment and medical record notes sent to mental health providers.
Arm/Group | CLASP Intervention | Safety Assessment and Follow up Evaluation
Number analyzed (Participants) | 18 | 30
score on a scale
  Baseline | 1.93 (0.68) | 1.98 (0.65)
  3 Month Followup | 1.30 (0.90) | 1.17 (0.84)
  6 Month Followup | 1.26 (0.84) | 1.23 (0.86)
  9 Month Followup | 0.93 (0.75) | 1.10 (0.86)
  12 Month Followup | 1.08 (0.90) | 1.06 (0.97)
Statistical Analysis 1: Comparison: CLASP Intervention vs Safety Assessment and Follow up Evaluation; Test type: Superiority; p = .49, RMANOVA — Adjusted for change in depression from baseline to 1yr (measured via QIDS); Partial eta squared = .02

4. Secondary Outcome: World Health Organization Disability Assessment Schedule (WHODAS) II
Description: The World Health Organization Disability Assessment Schedule (WHODAS II) is a validated, self-reported instrument assessing current impairment in functioning. Possible scores for each item range from 1 (None) to 5 (Extreme or cannot do). We calculated an Average Global Score for inclusion in analyses by dividing the total score by the number of items included in the measure (possible range of 1-5). Higher scores indicate greater impairment in functioning. We examined changes in overall functioning from baseline in these analyses.
Time Frame: Baseline, 3, 6, 9, & 12 month follow ups
Population: The number of participants in this analysis per group is smaller than was recruited at baseline due to dropout across time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CLASP Intervention | Safety Assessment and Follow up Evaluation
Number analyzed (Participants) | 17 | 30
score on a scale
  Baseline | 2.58 (0.55) | 2.54 (0.69)
  3 Month Followup | 2.12 (0.78) | 2.09 (0.79)
  6 Month Followup | 2.17 (0.72) | 2.07 (0.71)
  9 Month Followup | 2.00 (0.61) | 1.93 (0.76)
  1 Year Followup | 2.08 (0.82) | 2.04 (0.85)
Statistical Analysis 1: Comparison: CLASP Intervention vs Safety Assessment and Follow up Evaluation; Test type: Superiority; p = .96, RMANOVA — Adjusted for change in depression from baseline to 1yr (measured via QIDS); Partial eta-squared = .003

5. Secondary Outcome: Treatment History Interview
Description: We used an item measuring psychiatric hospitalizations from the Treatment History Interview to measure treatment utilization. Study participants indicated how many times they had been psychiatrically hospitalized since the prior study timepoint. We log transformed this variable at each timepoint to meet statistical assumptions of normality for our analyses.
Time Frame: 3, 6, 9, & 12 month follow up
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: log(psychiatric hospitalizations)
Arm/Group | CLASP Intervention | Safety Assessment and Follow up Evaluation
Number analyzed (Participants) | 23 | 32
log(psychiatric hospitalizations)
  3 Month Followup | 0.12 (0.20) | 0.07 (0.16)
  6 Month Followup | 0.03 (0.09) | 0.06 (0.14)
  9 Month Followup | 0.04 (0.10) | 0.06 (0.12)
  12 Month Followup | 0.05 (0.13) | 0.07 (0.14)
Statistical Analysis 1: Comparison: CLASP Intervention vs Safety Assessment and Follow up Evaluation; Test type: Superiority; p = .62, RMANOVA; Adjusted for change in depression from baseline to 1yr (measured via QIDS); Partial eta squared = 0.01

6. Secondary Outcome: Changes in Columbia Suicide Severity Rating Scale (C-SSRS) - Ideation Severity
Description: Intensity of ideation was measured using the Columbia Scale for Suicide Ideation intensity of ideation item. Item responses range from 1 (wish to be dead) to 5 (active suicidal ideation with specific plan and intent), with higher scores indicating more severe ideation. Minimum score on the ideation measure is 1 and maximum score is 5.
Time Frame: baseline, 3, 6, 9, & 12 month post-hospitalization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CLASP Intervention + Enhanced Monitoring | Safety Assessment and Follow up Evaluation + TAU
Number analyzed (Participants) | 25 | 32
units on a scale
  Baseline | 3.88 (0.73) | 4.16 (0.92)
  3 Month Followup | 2.56 (1.78) | 2.47 (1.81)
  6 Month Followup | 2.08 (1.91) | 1.66 (1.77)
  9 Month Followup | 1.64 (1.91) | 1.38 (1.74)
  12 Month Followup | 1.84 (1.89) | 1.25 (1.61)

ADVERSE EVENTS:
Time Frame: Adverse event data for each participant was collected for 12 months following baseline assessments.
Arm/Group | CLASP Intervention | Safety Assessment and Follow up Evaluation
All-Cause Mortality (participants affected / at risk) | 1/52 | 0/53
Serious Adverse Events (participants affected / at risk) | 21/52 | 17/53
Other Adverse Events (participants affected / at risk) | 0/52 | 0/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CLASP Intervention (N=52) | Safety Assessment and Follow up Evaluation (N=53)
Hospitalization for medical condition (Gastrointestinal disorders) | 1 (1) | 0 (0) — Pancreatitis
Hospitalization for suicide ideation or behavior (Psychiatric disorders) | 14 (19) | 9 (13) — Psychiatric hospitalization for suicide ideation or behavior
Hospitalization for substance use disorders (Psychiatric disorders) | 2 (4) | 4 (7) — Hospitalization for substance use disorder or detox
Hospitalization for chest pain (Cardiac disorders) | 1 (3) | 0 (0)
Hospitalization for excarbation of psychiatric symptoms (Psychiatric disorders) | 4 (7) | 6 (8) — Re-hospitalization for worsening of psychiatric symptoms such as PTSD or bipolar disorder
Hospitalization for pain (General disorders) | 2 (2) | 2 (2)
Medical hospitalization (General disorders) | 2 (2) | 0 (0) — broken bones/fractures

LIMITATIONS AND CAVEATS:
The dropout rate from baseline to the final timepoint (12 months) led to small numbers of subjects analyzed per group. Some completers had missing data for interim follow-up assessments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-03-31): https://cdn.clinicaltrials.gov/large-docs/41/NCT01894841/Prot_SAP_000.pdf
  • Informed Consent Form (2017-04-12): https://cdn.clinicaltrials.gov/large-docs/41/NCT01894841/ICF_001.pdf